CLINICAL TRIAL: NCT04117789
Title: Feasibility of Internet-delivered Cognitive Behavior Therapy for Adolescents With Mild to Moderate Depression: A Randomized Pilot Study Comparing Therapist-guided vs. Self-guided ICBT vs. Treatment as Usual
Brief Title: Feasibility of Internet-delivered CBT for Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Serlachius, PhD, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-03235
Record Dates: First submitted 2019-09-27; First posted 2019-10-07 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting post- and follow-up assessments will be blind to treatment allocation, for the full duration of the trial. The outcome measures are identical for both groups, ensuring that the assessors remain blind. At each follow-up assessment, participants will be reminded by their assessor to not reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation at each assessment point and motivate their choice. The blinding will be broken after the trial's final participant has finished his/her 3-month follow-up assessment (primary endpoint). The trial will end when the trial's final participant has finished his/her 3-month follow-up assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapist-guided ICBT for depression (Experimental): Participants will receive internet-delivered CBT with therapist support. The treatment consists of 8 online chapters with interactive features as videos and illustrations, delivered over a maximum of 10 weeks. The treatment has the main focus on behavioral activation.
  The adolescent and the caregiver are provided with their own separate programs and login to the treatment platform. The parent program also consists of eight chapters, including psychoeducation about depression and how to support their adolescent in treatment.
  The adolescents and caregivers have regular contact with a personal assigned therapist via written text messages in the platform. Participants are typically in contact with their therapist several times a week. The adolescent and caregiver can continue to access all treatment modules for the whole follow-up period (3 months), but without therapist-support.
  Interventions: Behavioral: Therapist-guided internet-delivered cognitive behavior therapy for depression in adolescents
- Self-guided ICBT for depression (Experimental): The self-guided ICBT for depression is identical to the therapist-guided ICBT intervention, however without the therapist support. To ensure patient-safety, there will be clear instructions to the patients and primary caregivers how to get in contact with the study team in case of acute problems, and there will be clinical routines to detect and manage deterioration or suicidal tendencies.
  Interventions: Behavioral: Self-guided internet-delivered cognitive behavior therapy for depression in adolescents
- Treatment as usual (TAU) (Active Comparator): Participants randomized to TAU, will be referred to the local CAMH's or primary care unit for children and youths and will be free to receive any treatment, either psychosocial, medical or the combination of both. The content of TAU and the treatment techniques used, will be monitored.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Therapist-guided internet-delivered cognitive behavior therapy for depression in adolescents — Participants will be assigned to a 10 weeks internet-delivered cognitive behavior therapy program with therapist support via an internet platform.
  Arms: Therapist-guided ICBT for depression
Behavioral: Self-guided internet-delivered cognitive behavior therapy for depression in adolescents — Participants will be assigned to a 10 weeks internet-delivered cognitive behavior therapy program without therapist support via an internet platform.
  Arms: Self-guided ICBT for depression
Other: Treatment as usual — Participants randomized to TAU, will be referred to the local CAMH's or primary care unit for children and youths and will be free to receive any treatment, either psychosocial, medical or the combination of both.
  Arms: Treatment as usual (TAU)

SUMMARY:
Prior to a properly powered randomized controlled study, evaluating efficacy and cost-effectiveness of ICBT, we will conduct a pilot study to investigate if the trial design is feasible, if therapist-guided and self-guided internet-delivered cognitive behavioral therapy (ICBT) is acceptable for adolescents with depression and to provide preliminary clinical efficacy data.

DETAILED DESCRIPTION:
A single-blind parallel-group pilot randomised controlled feasibility trial with the overall aim to develop two internet-delivered cognitive behaviour therapy interventions, therapist-guided and self-guided, for adolescents with mild to moderate Major Depressive Disorder (MDD) and their primary caregivers.

Patients can be either referred or self-referred. All potential participants are initially screened via telephone. This is followed by a face-to-face inclusion assessment. Participants who are eligible and have consented will be randomized into one of three trial arms; therapist-guided ICBT, self-guided ICBT or TAU. In the experimental arms, participants, e.g. the adolescent and at least one caregiver, either receive 10 weeks of therapist-guided or self-guided internet-delivered behavioural activation (BA). In the control arm, participants receive treatment as usual within the Child and Adolescent Mental Health Services (CAMHS) or primary care clinics. The primary endpoint will be at 3-month follow-up.

The primary objective is to evaluate the feasibility of the study design and trial procedures, including recruitment, withdrawal, drop out and attrition rates. The secondary objective is to (a) evaluate the acceptability of the ICBT interventions in regard to treatment satisfaction, credibility, reported adverse events, and program use, (b) to provide preliminary clinical efficacy data, and (c) to gather qualitative information on the experience of undergoing ICBT for depression from the perspective of adolescent patients, their caregivers and potential areas for improvement of future ICBT interventions.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of mild to moderate MDD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th ed.
* Willing to be randomized to either of the three treatment arms.
* Basic proficiency in Swedish, both adolescent and participating care-giver
* Regular access to a desktop or laptop computer connected to the internet, as well as a mobile phone to receive sms (one of each is enough per family).
* Stable medication with antidepressants, central stimulants and neuroleptics at least 6 weeks prior to inclusion.
* A minimum of one caregiver that is able to co-participate in the treatment.

Exclusion Criteria:

* Immediate risk to self or others, requiring urgent medical attention, such as suicidality, or repeated self-injurious behaviour.
* Other severe psychiatric disorders requiring other actions at first hand (e.g. diagnosis of organic brain disorder, intellectual disability, psychosis, bipolar disorder, eating disorder, or alcohol/substance dependence;
* Current social problems requiring other actions at first hand (e.g. bullying in school, abuse and/or neglect in the family; high and prolonged absence from school).
* Previous CBT for MDD within the last 12 months prior to assessment, for a minimum of 3 sessions other than psychoeducation with a qualified therapist within the 12 months prior to assessment.
* Current use of benzodiazepines.
* An ongoing psychological treatment for any other psychiatric disorder.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale - Revised (CDRS-R) | week 0, week 10, at 3 months follow-up
  CDRS-R is a semi-structured clinician interview, assessing level of depressive symptomatology. Total range is 17-113, with higher values representing a worse outcome. Change from baseline in depressive symptom severity on the CDRS-R at end of treatment, and at 3-months follow-up will be reported. Primary endpoint is 3 months follow-up.

SECONDARY OUTCOMES:
Treatment credibility and expectancy scale - adolescent and parent version | week 3
  This scale consists of four qualitative questions about treatment credibility, asking how well the treatment suits adolescents with depression, how much they believe this treatment will help him/her, if and to what extent they would recommend this treatment to a friend with depression and how much improvement they expect from the treatment. Total range is 4-20, with higher values representing higher credibility. Mean in total treatment credibility score on the "Treatment credibility scale" for each treatment group at week 3 will be reported.
The Client Satisfaction Questionnaire-8 (CSQ-8) - adolescent and parent version | week 10, at 3 months follow-up
  The CSQ-8 is an 8-item self-rated 4-point scale, measuring different aspects of satisfaction with treatment, e.g. perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction. Total range is 8 to 32, with higher values indicating higher satisfaction. Mean in total satisfaction scores on the CSQ-8 for each treatment group at end of treatment and at follow-up will be reported.
Need for further treatment - adolescent and parent version | week 10, at 3 months follow-up
  Investigate whether the participant considers her/himself in need of further treatment for her/his depression.
Negative Effects Questionnaire (NEQ-20) - adolescent and parent version | week 5, week 10, at 3 months-follow up
  NEQ-20 investigate participants' negative effects of psychological treatments. Total range is 0-80, with higher values representing a worse outcome.
  Descriptive data in negative effects of treatments on the NEQ-20 will be reported for participants randomized to either of the ICBT interventions at mid treatment, after end of treatment and at 3 months follow-up.
Treatment completion | week 10
  Adherence in terms of numbers of completed chapters for patients and their parents respectively in the ICBT interventions will be reported after 10 weeks. This data will be collected from the IT platform that delivers the ICBT interventions.
Therapist time | week 1 to week 10
  Total therapist time per patient an week will be reported for the ICBT interventions at the end of the pilot study. This data will be collected from the IT platform that delivers the ICBT interventions.
Clinical Global Impression Scale - Severity (CGI-S) | week 0, week 10, at 3 months follow-up
  CGI-S is developed to assess how mentally ill a specific patient compared to a particular patient population (e.g. with major depressive disorder) at a certain time.
  It consists of a single item rated on a seven-point scale ranging from 1="no symptoms" to 7="extreme symptoms". Change from baseline in global severity of depressive symptoms on the CGI-S at end of treatment, and at 3 months follow-up will be reported.
Clinical Global Impression - Improvement (CGI-I) | week 10, at 3 months follow-up
  CGI-I is developed to assess improvement of psychiatric symptoms for a specific patient compared to baseline. It consists of a single item rated on a seven-point scale ranging from 1="very much improved" to 7="very much worse". Change from baseline in global improvement of depressive symptoms to end of treatment and at 3 months follow-up on the CGI-I will be reported.
Children's global assessment scale (CGAS) | week 0, week 10, at 3 months follow-up
  The CGAS is a single item 1-100 scale that integrates psychological, social, and academic functioning in children as a measure of psychiatric disturbance. Higher values represent a worse outcome. Change from baseline in global functioning CGAS to end of treatment and at 3 months follow-up will be reported.
Short Mood and Feeling Questionnaire (SMFQ) - adolescent and parent version | week 0, weekly from week 1 to week 10, at 3 months follow-up
  The SMFQ is a 13-item self-reported measure of depressive symptoms. Total range is 0-26, with higher values representing a worse outcome. Change from baseline in adolescent- and parent-rated depressive symptoms on the SMFQ to week 10 and at 3 months follow-up, and weekly during treatment will be reported.
  Additionally, for this trial, we have also added a 14th item, aimed to assess suicide risk. This item is not included in the total score.
The Revised Children's Anxiety and Depression Scale, short (RCADS-S) -adolescent and parent version | week 0, week 10, 3 months follow-up
  The RCADS-S, a shortened version of the Spence Child Anxiety Scale, is a child and parent self-report measure of anxiety- and depression-related psychopathology. Only the anxiety subscales are administered in this study, since depressive symptoms are measured thoroughly by other measures. Total range is 0-45, with higher values representing a worse outcome. Change from baseline in adolescent- and parent-rated depressive symptoms on the RCADS-S to end of treatment and at 3 months follow-up will be reported.
Affective Reactivity Index (ARI) - adolescent and parent version | week 0, week 10, 3 months follow-up
  ARI is a parent- and self-rated measure of irritability and impairment due to irritability. Total range is 0-12, with higher values representing a worse outcome. Change from baseline in adolescent- and parent-rated irritability and impairment due to irritability on the ARI to end of treatment, and at 3-months follow-up will be reported.
Insomnia Severity Index (ISI) | week 0, week 10, at 3 months follow-up
  ISI, a brief screening measure of insomnia, a seven-item scale ranging from 0 to 28 points, with higher values representing a worse outcome. Change from baseline in sleep problems on ISI to end of treatment at 3 months follow-up will be reported.
Work and Social Adjustment Scale, youth version (WSAS-Y) - adolescent and parent version | week 0, week 10, 3 months follow-up
  WSAS-Y is a parent- and adolescent-rated scale of impaired functioning in school, everyday life, friends and social life, recreation and hobbies and family and close relationships. The scale generates a global score ranging from 0 to 40, with higher scores indicating greater impairment. Change from baseline in adolescent- and parent rated impairment and functioning on the WSAS-Y will be reported at the end of treatment, and at 3 months follow-up.
Working Alliance Inventory, Short (WAI-S) - adolescent and parent version | week 10, 3 months follow-up
  The WAI-S is scale measuring the participants perceived working alliance with their therapist. Total range 12-84, with higher scores indicating a better working alliance. Descriptive data on participants' perceived working alliance with their therapist, or with the program for participants in the self-guided ICBT, on the WAI-S will be reported at end of treatment and at 3-months follow up.
Kidscreen-10 Index - adolescent and parent version | week 0, week 10, at 3 months follow-up
  Kidscreen-10 assess the adolescents' general health-related quality of life. Total range from 10-50, with higher values indicating better health-related quality of life. Change from baseline in general health-related quality of life on the Kidscreen-10 will be reported at the end of treatment and at 3 months follow-up.

OTHER OUTCOMES:
Behavioral activation of Depression Scale - short form (BADS-S) | weekly during treatment (week 1 to week 10)
  The BADS-S is designed to track changes in proposed mediators of behavioral activation, e.g. activation and avoidance. Total range is from 0-54 with higher values indicating higher degree of activation and lower degree of avoidance.
  Changes during treatment in proposed mediators of behavioral activation on the BADS-S will be reported for the ICBT interventions.
Trimbos Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | week 0, week 10, at 3 months follow-up
  The TiC-P assess healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. In the present study no health economic evaluations will be conducted. Rather this instrument is included to gain feasibility data in preparation of a planned larger randomized controlled study. Therefore, no data on TiC-P will be reported in this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Child and Adolescent Psychiatry Research Center, Stockholm, Sweden

REFERENCES:
- [Derived] Andersson R, Vigerland S, Ahlen J, Widstrom H, Unger I, Serlachius E, Engberg H. "Therapy without a therapist?" The experiences of adolescents and their parents of online behavioural activation for depression with and without therapist support. Eur Child Adolesc Psychiatry. 2024 Jan;33(1):105-114. doi: 10.1007/s00787-023-02142-7. Epub 2023 Jan 17. PMID 36650254
- [Derived] Grudin R, Ahlen J, Mataix-Cols D, Lenhard F, Henje E, Mansson C, Sahlin H, Beckman M, Serlachius E, Vigerland S. Therapist-guided and self-guided internet-delivered behavioural activation for adolescents with depression: a randomised feasibility trial. BMJ Open. 2022 Dec 26;12(12):e066357. doi: 10.1136/bmjopen-2022-066357. PMID 36572500